CLINICAL TRIAL: NCT01469442
Title: Postoperative Biliary Fistula Prevention After Hepatectomy by External Biliary Duct Stent:Prospective Multicenter Randomized Trial
Brief Title: Postoperative Biliary Fistula Prevention After Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08 114 01
Record Dates: First submitted 2011-07-04; First posted 2011-11-10 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Hepatectomy
Keywords: Biliary fistula; prevention; hepatectomy; external stent; Hepatectomy of more 2 segments; Not emergency or laparoscopy surgery
MeSH Terms: conditions — Biliary Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- external biliary duct stent (Experimental): 'External Biliary duct stent in the bile duct by cystic way'
  Interventions: Procedure: External Biliary duct stent in the bile duct by cystic way
- without external biliary duct stent (No Intervention)

INTERVENTIONS:
Procedure: External Biliary duct stent in the bile duct by cystic way — The size of the external biliary duct stent depending of cystic duct size
  Arms: external biliary duct stent

SUMMARY:
Aim : Effect of external biliary duct stent after hepatectomy on the occurence of postoperative biliary fistula.

Methods : French prospective multicenter randomized trial. Population study: Adult patients who underwent hepatectomy (> 2 segments) on non-cirrhotic liver.

Hypothesis: decreased postoperative biliary fistula from 15% to 5% with the presence of a external biliary duct stent. With this hypothesis, the number of patients required to be equal to 152 per group for a total of 304 patients.

Outcome measure: Primary : Postoperative biliary complications (biliary fistula, biloma, biliary peritonitis) Secondary : All morbidity, mortality, additional manoeuvres to treat biliary fistula, during of hospital stay and biliary fistula.

Follow up: A follow-up of patients 3 months after surgery for all patients. The planned total duration of the study is 3 years and 3 months.

DETAILED DESCRIPTION:
After performing the hepatectomy and verification of hemostasis, patients were randomized (external biliary duct stent or not) by sealed envelopes. Systematic intraoperative test with methylene blue or air by the external biliary duct stent (EBDS) will necessary for all patients. Intra-abdominal drainage or not and type will be at the discretion of the surgeon. The EBDS will be left open for the first 7 postoperative days and then clamped. The EBDS will be removed during a consultation 5 weeks after surgery. Both groups of patients will be reviewed at 3 months after surgery, it will be noted at this point the possible complications related to the presence of EBDS (leakage from the drain, drop..). If patients are hospitalized more than five weeks, the study will stop at their consultation three months or the day of the consultation where the DTC is removed if it is still present at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given his informed consent and signed consent
* Hepatectomy at least 2 segments of liver parenchyma for a benign or malignant disease by laparotomy
* Not cirrhotic liver

Exclusion Criteria:

* Surgery made in emergency
* Surgery by laparoscopy
* Need to draw up a bilic-digestive anastomosis
* Liver cirrhosis
* History of cholecystectomy
* Resection of less than 2 segments
* Preoperative jaundice (total bilirubin> 30 micromol / l)
* Presence of preoperative biliary drainage
* Patients requiring the installation of a drain transcystic during the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Postoperative biliary fistula | 3 months after surgey
  3 forms of diagnosis : bile in the intra-abdominal drainage; presence of an intra-abdominal collection of bile liquid (biloma); presence of an effusion of bile in the abdominal space (biliary peritonitis).

SECONDARY OUTCOMES:
Morbidity | 3 months after surgey
  additional maneuvers for treat biliary fistula, during of hospital stay, during of biliary fistula
Mortality | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice MUSCARI, MD, Principal Investigator — University Hospital, Toulouse
Locations (12):
- France (12):
  - CHU, Amiens
  - Hotel Dieu, Clermont-Ferrand
  - Hôpital beaujon, Clichy
  - Hôpital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU la conception, Marseille
  - Hôpital St Eloi, Montpellier
  - Hotel Dieu, Nantes
  - Hôpital Saint Antoine, Paris
  - hôpital Haute Pierre, Strasbourg
  - Toulouse Purpan, Toulouse
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maulat C, Regimbeau JM, Buc E, Boleslawski E, Belghiti J, Hardwigsen J, Vibert E, Delpero JR, Tournay E, Arnaud C, Suc B, Pessaux P, Muscari F. Prevention of biliary fistula after partial hepatectomy by transcystic biliary drainage: randomized clinical trial. Br J Surg. 2020 Jun;107(7):824-831. doi: 10.1002/bjs.11405. Epub 2020 Jan 9. PMID 31916605